CLINICAL TRIAL: NCT00440882
Title: Changes of Transforming Growth Factor b1 and Procollagen III in Patients With Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Dr FOREL JM, Assistance Publique Hopitaux De Marseille
Other Study IDs: 2004/16
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-10

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Transforming Growth Factor-b1 (TGF-b1) is involved in the development of acute lung injury and in the fibroproliferation during acute respiratory distress syndrome (ARDS). Procollagen III Peptide (PIIINP) is a validated marker of fibroproliferation. PIIINP is associated with death in ARDS patients. The simultaneous changes of TGF-b1 and PIIINP were never studied in patients with ARDS. The relationships between TGF-b1 and the outcome of ARDS are unknown.

The aim of the study is to analyse the changes of TGF-b1 and PIIINP during ARDS and to show the relationships between TGF-b1 - PIIINP and the outcomes of ARDS.

DETAILED DESCRIPTION:
Primary outcome: To analyse the changes of Transforming Growth Factor b1 and Procollagen III during the acute respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

* ARDS with a PaO2/FIO2 < 200 mmHg at a positive end-expiratory pressure (PEEP) ³ 5 cm H2O
* ARDS criteria from less than 24 hours
* Informed consent

Exclusion Criteria:

* Pregnancy
* Chronic interstitial or fibrosis lung diseases
* Hepatic chronic disease
* Neutropenia £1 G/l
* Corticosteroid (more than 200 mg/day of hydrocortisone or equivalent, less than 2 weeks before inclusion)
* Immunosuppressive therapy within the last 30 days
* Participation in any investigational drug or devices study within 30 days prior study entry

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients whom suffered ARDS with a PaO2/FIO2 < 200 mmHg at a positive end-expiratory pressure (PEEP) ³ 5 cm H2O and for which ARDS criteria from less than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie FOREL, MD, Principal Investigator — AP-HM
Locations (1):
- Hopital Sainte Marguerite, Marseille, France